CLINICAL TRIAL: NCT07033117
Title: The RaDIANT Health Systems Intervention for Improving Access to Kidney Transplantation
Brief Title: RaDIANT Health Systems Intervention
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Indiana University Health (Other); Emory Healthcare (Other); Piedmont Healthcare (Other); Medical University of South Carolina (Other); Duke University (Other)
Responsible Party: Principal Investigator, Rachel Patzer, PhD, MPH, Professor, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 18998 - Aim 2; R01DK136283 (NIH)
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: End Stage Renal Disease (ESRD); Kidney Disease
MeSH Terms: conditions — Kidney Failure, Chronic; Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multi-Component Intervention (Experimental): Five participating transplant centers will multicomponent intervention in their management of patients referred to their transplant center for a kidney transplantation. The intervention will consist of: (1) required performance feedback reports on closed referrals; and a set of optional components that may be implemented variably by centers, including; (2) contacting patients via their preferred method; (3) phone calls to the dialysis facility during the patient's dialysis session; (4) phone calls to the referring or other provider; (5) use of a multi-module, secure, web-enabled software application called Transplant Referral EXchange (T-REX) or secure email to communicate patient status and no-show information; and (6) communication tracking and audit. Dialysis facilities in GA, NC, SC, and IN will receive resources to support an awareness campaign to support implementation of intervention activities within transplant centers.
  Interventions: Other: Performance Feedback Reports on Referral and Evaluation Closures; Other: Dialysis Facility Awareness Campaign; Other: Patient Contact via Preferred Method; Other: Phone Call to Dialysis Facility During the Patient's Dialysis Session; Other: Phone Call to Provider; Other: Transplant Referral Communication Platforms or Email to Communicate Patient Status and No-Show; Other: Audit and Tracking of Patient Contact Attempts Prior to Referral Closure

INTERVENTIONS:
Other: Performance Feedback Reports on Referral and Evaluation Closures — Performance feedback reports will reflect each transplant center's performance related to kidney transplant evaluation initiation and referral closure. These reports aim to help centers understand common reasons why patients do not initiate the evaluation process or failed to proceed beyond the evaluation process, and to identify patterns in referral and evaluation closure practices. Reports will be individualized and distributed quarterly to the transplant center champion by the intervention lead.
Other: Dialysis Facility Awareness Campaign — As part of the intervention, dialysis centers will participate in an Awareness Campaign designed to educate staff about transplant center quality improvement efforts and how they may be contacted as part of the project. This campaign may include brief webinars or informative documents distributed via platforms such as IPRO Learn.
Other: Patient Contact via Preferred Method — Transplant centers will contact patients using their preferred method of communication.
Other: Phone Call to Dialysis Facility During the Patient's Dialysis Session — Facilities will enhance their patient communication procedures by making a phone call to the dialysis facility during the patient's dialysis session if the patient has not responded to initial outreach attempts. This additional step increases the likelihood of reaching the patient during a time when they are accessible and can engage in scheduling or follow-up.
Other: Phone Call to Provider — Transplant centers will enhance their outreach procedures by making a phone call to the referring provider (e.g., nephrologist, medical assistant) or another provider involved in the patient's care (e.g., primary care provider) in the event of self-referral if the patient has not responded to initial outreach attempts or "no-shows" an initial evaluation appointment. This additional step ensures that the referring provider is informed of the patient's progress and can assist in re-engagement or decision-making prior to referral closure.
Other: Transplant Referral Communication Platforms or Email to Communicate Patient Status and No-Show — Transplant center staff will utilize transplant referral communication platforms and/or email to communicate updates to dialysis staff regarding patient status (e.g., unable to contact the patient or no-show) before referral closure.
Other: Audit and Tracking of Patient Contact Attempts Prior to Referral Closure — Transplant center staff will continue internally tracking the frequency that a patient is contacted before closure and the date of closure, in alignment with center standard practice. This intervention introduces an audit process to be conducted before closure to ensure that all contact attempts (including one or more attempts to contact the patient directly, one or more phone calls to the alternate preferred contact, or one or more attempted contacts to the dialysis unit to connect with the patient), in alignment with center communication procedures, are appropriately executed.

SUMMARY:
The overarching goal of the proposed study is to determine whether the addition of structural interventions at the health system level targeting upstream barriers in the transplant process will improve access to transplant evaluation start.

ELIGIBILITY:
Inclusion Criteria:

* Five large transplant centers (Emory Transplant Center and Piedmont Transplant Center in Atlanta, GA; Medical University of SC; Duke University in Durham, NC; and Indiana University in Indianapolis, IN) ~800 referring dialysis center referring to these transplant centers

Exclusion Criteria:

* Individuals referred, initiating evaluation, and waitlisted at non-participating start centers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14000 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in transplant evaluation start within 6 months of transplant referral | Baseline, Post Intervention (Up to one year)
  The difference in the proportion of patients starting transplant evaluation within 6 months of being referred from baseline to up to one-year post-intervention

SECONDARY OUTCOMES:
Change in transplant waitlisting | Baseline, Post Intervention (Up to one year)
  The difference in the proportion of patients waitlisted from baseline and up to one-year post-intervention
Change in transplant receipt among those who were waitlisted | Baseline, Post Intervention (Up to one year)
  The difference in the proportion of patients who received a transplant among those who were waitlisted from baseline and up to one-year post-intervention

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Piedmont Transplant Institute, Atlanta, Georgia
  - Emory Transplant Center, Atlanta, Georgia
  - IU Health Transplant - Indianapolis, Indianapolis, Indiana
  - Duke Transplant Center, Durham, North Carolina
  - MUSC Mid-Carolinas Transplant Center, Lancaster, South Carolina

IPD SHARING:
Plan to Share IPD: No